CLINICAL TRIAL: NCT00451802
Title: A Pilot Scheme - Specimen Collection of Health Management Center
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9261701410; NTUH93A07; NTUH94A02
Record Dates: First submitted 2007-03-22; First posted 2007-03-26 (Estimated); Last update posted 2007-03-26 (Estimated); Status verified 2005-01

CONDITIONS: Healthy
Keywords: Biotechnology; Specimen; Health Management Center

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other

SUMMARY:
Biomedical and biotechnology industry is internationally regarded as the most brilliant star performer of the future. The development of biomedical depends on a high quality academic research environment, while innovation and uniqueness should be emphasized for the development of biotechnology industry. The successful development of biotechnology industry will be impossible if the development is not based on extensive and in-depth research work and verification acquired from clinical implementation. Based on these concepts, the resources of research materials, especial of human being, are going to be essential. Thus, a programmable and systematic collection of clinical specimen would become one of the potential properties in hospital. This is a two-year pilot scheme, and was designed to start collecting specimen from "Health Management Center" in NTUH. This pilot scheme will address important issues of manpower, finances, and data merging for evaluation of biotechnological related specimen collection, such as cell or tissue bank, in the future.

DETAILED DESCRIPTION:
Biomedical and biotechnology industry is internationally regarded as the most brilliant star performer of the future. The development of biomedical depends on a high quality academic research environment, while innovation and uniqueness should be emphasized for the development of biotechnology industry. The successful development of biotechnology industry will be impossible if the development is not based on extensive and in-depth research work and verification acquired from clinical implementation. Based on these concepts, the resources of research materials, especial of human being, are going to be essential. Thus, a programmable and systematic collection of clinical specimen would become one of the potential properties in hospital. This is a two-year pilot scheme, and was designed to start collecting specimen from "Health Management Center" in NTUH. This pilot scheme will address important issues of manpower, finances, and data merging for evaluation of biotechnological related specimen collection, such as cell or tissue bank, in the future.

There are 12471 persons who take the health examination in Health Management Center during 2004 Mar -2005 Dec. Subjects agree to be invovled in the study asre assigned as "respondent". For those who disgree to be involved in the study are assigned as "non-respondent". There are 6261 respondents and 6210 non-respondents in this study. 63% of respondents and 51% of non-respondents are males. There is a lower distribution in smoking, history of hypertension, and history of hyperlipidemia in respondents than in non-respondents. Respondents have lower level of triglyceride, HDL, LDL in blood than non-respondents do.

ELIGIBILITY:
Inclusion Criteria:

* Biotechnology
* Persons who take the health examination in Health Management Center during 2004 Mar - 2005 Dec.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 7000
Dates: Start 2003-01; Study Completion 2005-12

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Fong Chen, MD. PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- Chen Ming-Fong, Taipei, Taiwan